CLINICAL TRIAL: NCT04494347
Title: Watchman for Patients With Atrial Fibrillation Undergoing Transcatheter Mitral Valve Repair (WATCH-TMVR)
Acronym: WATCH-TMVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mohamad Adnan Alkhouli, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-010047
Record Dates: First submitted 2020-07-01; First posted 2020-07-31 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Nonvalvular Atrial Fibrillation; Severe Degenerative Mitral Regurgitation

STUDY DESIGN:
Intervention Model Description: This is a prospective multicenter registry of 25 patients who are planned to undergo TMVr with MitraClip and also have an indication for LAAO with the commercially available WATCHMAN device. All patients will undergo TMVr first under general anesthesia and transesophageal echo (TEE) guidance. At the conclusion of the TMVr procedure, the patient will undergo LAAO with the Watchman device using the same transseptal access the was obtained to perform the TMVr. Patients will receive oral anticoagulation with warfarin (or a direct anticoagulant) and subsequent antiplatelet therapy as per standard of care and outlined in protocol for 6 weeks. After 6 weeks, patients will have TEE done as per standard of care in addition to office visit and complete clinical and neurological evaluation. Continuation or discontinuation of oral anticoagulation will depend on the 45-day TEE findings. The anticipated duration of the Clinical Investigation will be 12 months.
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): This is not a randomized study. Patients who are clinically indicated for both procedures will be offered the option to enroll in this registry for a combined procedure. Otherwise, they will undergo TMVr and LAAO in two separate session as clinically indicated (standard of care).
  Interventions: Procedure: MitraClip TMVR and Watchman LAAO

INTERVENTIONS:
Procedure: MitraClip TMVR and Watchman LAAO — The MitraClip device is a percutaneous edge-to-edge repair device that is intended to approximate the anterior and posterior mitral valve leaflets in patients with severe symptomatic mitral regurgitation with suitable anatomy. Device versions/types: MitraClip NTr, MitraClip XTr. The WATCHMAN device is a self-expanding left atrial appendage occlusion (LAAO) device with a porous covering on the proximal face. Device sizes: 21 mm, 24 mm, 27 mm, 30 mm, 33 mm.

SUMMARY:
WATCH-TMVR (Watchman for Patients with Atrial Fibrillation Undergoing Transcatheter Mitral Valve) Clinical Trial have the main objective to assess the feasibility of combining clinically indicated MitraClip TMVR and Watchman LAAO in one setting.Mayo Clinic will be the data coordinating center for this trial, which will include up to 3 sites.

DETAILED DESCRIPTION:
Left atrial appendage closure using the Watchman device procedure is approved by the FDA for patients with nonvalvular atrial fibrillation who have an indication for oral anticoagulation to reduce stroke risk but who also have a rational to seek an alternative to long-term anticoagulation (e.g., recurrent bleeding, fall risk). Transcatheter mitral valve repair with the MitraClip device is approved by the FDA for patients with severe degenerative mitral regurgitation who are deemed to be at high-risk for valve surgery and patients with severe secondary MR despite optimal medical therapy. It is also anticipated that the device will soon be approved for patients with severe symptomatic functional mitral regurgitation based on the results of the COAPT trials. Atrial fibrillation is common in patients referred for TMVr. A recent study from the Mayo Clinic documented that up to 50% of patients undergoing TMVr might qualify for LAA based on their risk assessment. Both procedures are performed via a large bore femoral venous access, and utilize transseptal puncture, general anesthesia, and transesophageal echo guidance. Hence, combining the two procedures in one session might provide incremental benefit to those patients by avoiding the risk of repeated large-bore access, transseptal puncture, and general anesthesia. A limited number of case reports illustrated the safety and feasibility of a combined TMVr with LAAO when clinically indicated. Experience with combined TMVr/LAAO in the United States is limited, mostly due to the lack of supportive data and concerns about the incremental cost of the Watchman device that might not be covered by the Center for Medicare Services (CMS) per current guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women ≥ 18 years of age;
2. The patient has severe symptomatic mitral regurgitation meet criteria for the commercially available MitraClip;
3. The patient also has documented paroxysmal, persistent, or permanent atrial fibrillation AND The patient meets the WATCHMAN labeling guidelines;
4. The patient is eligible for short-term oral anticoagulation therapy with Warfarin or a direct oral anticoagulant;
5. The patient or legal representative is able to understand and willing to provide written informed consent to participate in the trial;
6. The patient is able and willing to return for required follow-up visits.

Exclusion Criteria:

1. Mitral valve anatomy not deemed suitable for TMVr;
2. Moderate to severe mitral stenosis (mean gradient >10 mmHg or MVA <1.5 cm2);
3. Contraindication for short-term anticoagulation;
4. The patient has intra-cardiac thrombus as visualized by TEE within 1 week prior to Watchman procedure;
5. Prior occlusion of LAA;
6. Implanted mechanical mitral valve;
7. The patient requires long-term warfarin therapy due to:

   1. Secondary to conditions such as prior arterial embolism or other indications such as pulmonary embolism or deep vein thrombosis within the previous 6 months.
   2. The patient is in a hypercoagulable state.
8. Exclude the patient if per medical record documentation the patient meets any of the following criteria: • Thrombosis occurring at under 40 years age • Idiopathic or recurrent VTE (venous thromboembolism • Thrombosis at an unusual site (cerebral veins, hepatic veins, renal veins, IVC, mesenteric veins) • Family history of VTE or of inherited prothrombotic disorder, recurrence/extension of thrombosis while adequately anti-coagulated;
9. The patient is actively enrolled in another trial of a cardiovascular device or an investigational drug (post-market study and registries are acceptable);
10. The patient is pregnant, or pregnancy is planned during the course of the investigation if patient is of child bearing potential;
11. Any clinically significant medical condition or presence of any laboratory abnormality performed prior to randomization that is considered by the investigator to be clinically important and could interfere with the conduct of the study or not meeting procedure guidelines for WATCHMAN or TMVr with MitraClip;
12. The patient has a life expectancy of less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality rate | 45 days post procedure
  Total number of Subject's Death
All-cause mortality rate | 1 Year post procedure
  Total number of Subject's Death
Serious Adverse Events (SAEs) | 45 days post procedure
  Total number of Subject's experiencing SAEs such Stroke, life-threatening or major bleeding.
Serious Adverse Events (SAEs) | 1 Year post procedure
  Total number of Subject's experiencing SAEs such Stroke, life-threatening or major bleeding.

SECONDARY OUTCOMES:
SAEs related to the Study devices | 1 Year
  Total number of the Subject's to experience SAEs as related to Watchman and the LAAO devices.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Adnan (Mohamad) Alkhouli, MD, Principal Investigator — Mayo Clinic
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials